CLINICAL TRIAL: NCT05842213
Title: Randomized, Double-blind, 2-arm Multicenter Study to Investigate the Efficacy, Safety and Immunogenicity Between Subcutaneous AVT05 and EU-approved Simponi® in Subjects with Moderate to Severe Rheumatoid Arthritis
Brief Title: Comparative, Multicenter Study in Subjects with Rheumatoid Arthritis, ALVOFLEX
Acronym: ALVOFLEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVT05-GL-C01
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AVT05 (Experimental): AVT05 is the proposed biosimilar to Simponi. Subjects in this arm will receive AVT05 50mg s.c. every 4 weeks until week 48.
  Intervention: Biological: Golimumab
  Interventions: Biological: AVT05 (proposed biosimilar to golimumab)
- Simponi (Active Comparator): Subjects in this arm will receive EU Simponi 50mg s.c. every 4 weeks until week 12. At week 16 responders will be re-randomized in a 1:1 ratio to receive either:
  AVT05 50mg s.c. every 4 weeks until week 48 Simponi 50mg s.c. every 4 weeks until week 48 Intervention: Biological: Golimumab
  Interventions: Biological: AVT05 (proposed biosimilar to golimumab); Biological: Simponi (Golimumab)

INTERVENTIONS:
Biological: AVT05 (proposed biosimilar to golimumab) — AVT05 is a recombinant human IgG1қ mAb developed as a subcutaneous injection
Biological: Simponi (Golimumab) — Simponi (Golimumab) is a recombinant human IgG1қ mAb developed as a subcutaneous injection
  Arms: Simponi

SUMMARY:
This is a study to compare the efficacy, safety and immunogenicity of AVT05 versus EU-Simponi® in combination with methotrexate (MTX) in subjects with moderate to severe rheumatoid arthritis (RA).

The study will consist of up to 4-week Screening Period, a 48-week Treatment Period, and a 4-week Safety Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with active RA according to ACR/EULAR 2010 classification criteria
* Subjects diagnosed with moderately to severe active RA as defined by ≥ 6 swollen (out of 66) and ≥6 tender (out of 68) joint counts, CRP >1mg/l and with at least one of positive rheumatoid factor, positive anti-citrullinated peptide antibodies and/or evidence of 1 joint erosion of hands, wrist of dominant hand or feet at screening
* Subjects must have taken methotrexate for ≥12 weeks

Exclusion Criteria:

* Prior treatment with biologics or Janus kinase inhibitors that may be used as disease-modifying anti-rheumatic drugs
* Any past or concurrent medical conditions that could potentially increase the subject's risks or that would interfere with the study evaluation, procedures or study completion
* Major chronic inflammatory disease or connective tissue disease other than RA or any active autoimmune disease
* Presence of chronic obstructive pulmonary disease
* Presence of chronic heart failure NYHA class III or IV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Demonstrate comparative efficacy of AVT05 with EU-approved Simponi as measured by DAS28-CRP at week 16. | Week 16
  Change from baseline in DAS28-CRP response criteria at week 16

SECONDARY OUTCOMES:
Assess additional efficacy measures of AVT05 and EU-Simponi in terms of DAS28-CRP | Weeks 4, 8, 12, 24, 32, 40, 48 and 52
  Change from baseline in DAS28-CRP response criteria at weeks 4, 8, 12, 24, 32, 40, 48 and 52
Assess additional efficacy measures of AVT05 and EU-Simponi in terms of ACR20/50/70 and its individual components throughout the study | Weeks 4, 8, 12, 16, 24, 32, 40, 48 and 52
  Percentage of subjects achieving ACR20/50/70 at weeks 4, 8, 12, 16, 24, 32, 40, 48 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bucknall, Study Director — Alvotech Swiss AG
Locations (1):
- Rheumatology clinic, University Multiprofile Hospital for Active Treatment Kaspela, Plovdiv, Bulgaria

REFERENCES:
- [Derived] Luque M, Zhelyazkova K, Vashishta L, Rai M, Sattar A, Petrovic K, Bucknall R, Leutz S, Berti F. Efficacy and Safety of Biosimilar AVT05 Versus Reference Product Golimumab in Combination with Methotrexate in Moderate-to-Severe Rheumatoid Arthritis: 52-Week Results of a Randomized, Parallel-Group, Double-Blind Study. BioDrugs. 2025 Nov 3. doi: 10.1007/s40259-025-00748-8. Online ahead of print. PMID 41182658